CLINICAL TRIAL: NCT02180659
Title: A Randomized, Double-Blind, Double-Dummy, Active-Controlled Multicenter Study of Adult Outpatients With Opioid Dependence Transitioned From a Daily Maintenance Dose of 8 mg or Less of Sublingual Buprenorphine or Buprenorphine/Naloxone to Four Probuphine® Subdermal Implants
Brief Title: A Study of Adult Outpatients With Opioid Dependence Transitioned From a Daily SL Buprenorphine to Probuphine® Subdermal Implants
Acronym: PRO-814
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Titan Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRO-814
Record Dates: First submitted 2014-07-01; First posted 2014-07-03 (Estimated); Results first posted 2018-12-05 (Actual); Last update posted 2019-01-11 (Actual); Status verified 2018-11

CONDITIONS: Opioid Dependence
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Buprenorphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- buprenorphine implants + placebo tablets (Experimental): Four 80 mg Probuphine implants + daily SL placebo tablets
  Interventions: Drug: Buprenorphine implant; Drug: sublingual placebo tablets
- buprenorphine tablets + placebo implants (Active Comparator): Daily SL BPN tablets (≤8 mg/daily) + four placebo implants
  Interventions: Drug: sublingual buprenorphine tablets; Drug: placebo implants

INTERVENTIONS:
Drug: sublingual buprenorphine tablets
  Arms: buprenorphine tablets + placebo implants
Drug: Buprenorphine implant
  Arms: buprenorphine implants + placebo tablets
Drug: placebo implants
  Arms: buprenorphine tablets + placebo implants
Drug: sublingual placebo tablets
  Arms: buprenorphine implants + placebo tablets

SUMMARY:
The primary objective of the study is to demonstrate maintenance of treatment efficacy when transferring adult outpatients with opioid dependence, who are clinically stabilized on 8 mg or less of sublingual (SL) buprenorphine (BPN), to 4 Probuphine implants compared to SL BPN.

The secondary objective of the study is to confirm safety of 4 Probuphine implants in adult outpatients with opioid dependence who are clinically stabilized on 8 mg or less of SL BPN.

DETAILED DESCRIPTION:
This is a randomized, double-blind, double-dummy, active-controlled multi-center study to evaluate the efficacy of transition to four 80 mg Probuphine implants in adult outpatients with opioid dependence, who are clinically stabilized on 8 mg or less of SL BPN. The study will include 3 Phases; Screening, Maintenance and Follow-up.

Medical and eligibility screening should occur within 2 weeks of the first Maintenance Phase visit. The Screening Visit will include standard medical screening procedures, complete medical/psychosocial history, urine toxicology and detailed substance use and treatment history.

All subjects who have provided written informed consent and have met the other study entry criteria will be eligible for randomization. Following confirmation of eligibility, subjects will be randomized to one of two treatment groups in a 1:1 ratio:

* Treatment Group A: Daily SL BPN tablets (≤8 mg/daily) + four placebo implants
* Treatment Group B: Four 80 mg Probuphine implants + daily SL placebo tablets

Implants will be surgically inserted on Day 1 (Baseline and Initiation of Study Drugs Visit). On Post-Implant Visit, additional follow-up safety and implant assessment procedures will be conducted. Subjects will return for monthly study visits on Weeks 4, 8, 12, 16, 20, and 24 (End of Treatment Visit). In addition to the monthly scheduled visits, subjects will provide 4 random urine toxicology samples throughout the 24-week treatment period.

A total of 10 urine toxicology samples will be collected; 6 at scheduled visits (1 per month) and 4 at random urine toxicology visits throughout the 24-week treatment period. At the scheduled visits, other assessments of efficacy and safety will be collected. Implants will be removed at the End of Treatment Visit on Week 24.

Following Week 24, subjects will be re-transitioned back to usual care (pre-trial), as needed. During Week 25, telephone contact will be made with all subjects. and Week 26 will include an on-site visit to the clinic for final follow-up assessments (Follow-up Visit).

ELIGIBILITY:
Inclusion Criteria:

1. Subject must provide written informed consent prior to the conduct of any study-related procedures.
2. Male or female, 18-65 years of age, inclusive.
3. Primary diagnosis of opioid dependence (DSM-IV-TR).
4. Subject is considered clinically stable by their treating healthcare provider and confirmed by the following:

   1. Subject must be on SL BPN treatment for at least 6 months.
   2. Subject must have been on a SL BPN dose of 8 mg or less daily for at least the last 90 days prior to Screening.
   3. No positive urine toxicology results for illicit opioids in the last 90 days.
5. Free from significant withdrawal symptoms (score of ≤ 5 on the Clinical Opiate Withdrawal Scale [COWS]), as measured at the Screening Visit.
6. Female subjects of childbearing potential must be willing to use a reliable method of contraception during the entire study (Screening Visit to Follow-Up Visit).

Exclusion Criteria:

1. Current diagnosis of Acquired Immune Deficiency Syndrome (AIDS).
2. Current diagnosis of chronic pain syndrome requiring chronic opioid treatment, or conditions associated with acute episodic flares that require opioid treatment.
3. Pregnant or lactating or planning to become pregnant during the study.
4. Hypersensitivity or allergy to ethylene vinyl acetate (EVA)-containing substances or naloxone.
5. Recent scarring or tattoos on their upper arms, or a history of keloid scarring.
6. Requires current use of agents metabolized through CYP 3A4 such as azole antifungals (e.g., ketoconazole), macrolide antibiotics (e.g., erythromycin), or protease inhibitors (e.g., ritonavir, indinavir, and saquinavir).
7. History of coagulopathy within the past 90 days, and/or current anti-coagulant therapy such as warfarin.
8. Current DSM-IV-TR diagnosis for substance dependence on any other psychoactive substances other than opioids or nicotine (e.g., alcohol, cocaine).
9. Significant symptoms or other factors which in the opinion of the Investigator would preclude compliance with the protocol, subject safety, adequate cooperation in the study, or obtaining informed consent.
10. Current medical conditions such as severe respiratory insufficiency that may prevent the subject from safely participating in study.
11. Any pending legal action that could prohibit participation or compliance in the study.
12. Exposure to any investigational drug within the 8 weeks prior to Screening.
13. Aspartate aminotransferase levels ≥3 X the upper limit of normal, alanine aminotransferase levels ≥ 3 X the upper limit of normal, total bilirubin ≥ 1.5 X the upper limit of normal, or creatinine ≥ 1.5 X upper limit of normal on the Screening laboratory assessments.
14. Clinically significant low platelet count on the Screening laboratory assessments, according to the Investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 177 (Actual)
Dates: Start 2014-07; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

REFERENCES:
- [Derived] Rosenthal RN, Lofwall MR, Kim S, Chen M, Beebe KL, Vocci FJ; PRO-814 Study Group. Effect of Buprenorphine Implants on Illicit Opioid Use Among Abstinent Adults With Opioid Dependence Treated With Sublingual Buprenorphine: A Randomized Clinical Trial. JAMA. 2016 Jul 19;316(3):282-90. doi: 10.1001/jama.2016.9382. PMID 27434441

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient enrolled: 26 June 2014. Last patient completed: 18 May 2015
  A total of 21 Investigators participated in the study, across 21 sites in the United States.
Pre-assignment Details: 211 patient were screened and of those,177 subjects were enrolled and randomized into the study.
Groups:
- Buprenorphine Implants + Placebo Tablets: Four 80 mg Probuphine implants + daily SL placebo tablets
  Buprenorphine implant
  sublingual placebo tablets
- Buprenorphine Tablets + Placebo Implants: Daily SL BPN tablets (≤8 mg/daily) + four placebo implants
  sublingual buprenorphine tablets
  placebo implants
Period: Overall Study
Arm/Group | Buprenorphine Implants + Placebo Tablets | Buprenorphine Tablets + Placebo Implants
Started | 87 | 89 (N=90 randomized, however N=89 received study medication)
Completed | 81 | 84
Not Completed | 6 | 5
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 4 | 2
Not completed — Subject incarcerated during conduct | 1 | 0
Not completed — Withdrawal by Subject | 0 | 2
Not completed — AT REQUEST OF THE SPONSOR | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Buprenorphine Implants + Placebo Tablets | Buprenorphine Tablets + Placebo Implants | Total
Number analyzed (Participants) | 87 | 89 | 176
Age, Continuous [Mean (Full Range); unit: Years] | 38 [21 to 63.0] | 39 [22 to 64.0] | 39 [21 to 64.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 37 | 72
  Male | 52 | 52 | 104
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 6
  Not Hispanic or Latino | 84 | 86 | 170
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 3 | 2 | 5
  White | 82 | 85 | 167
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
BMI [Mean (Full Range); unit: kg/m^2] | 28 [14 to 46.4] | 27 [19 to 50.6] | 28 [14 to 50.6]
Primary opioid of abuse [Count of Participants; unit: Participants]
  Prescription opioid pain reliever | 66 | 65 | 131
  Heroin | 15 | 22 | 37
  Other | 5 | 2 | 7
  Not reported | 1 | 0 | 1
Time since first opioid abuse [Mean (Full Range); unit: Years] | 11.2 [1.4 to 36.6] | 11.5 [1.6 to 45.6] | 11.3 [1.4 to 45.6]
Time from first diagnosis of opioid dependence [Mean (Full Range); unit: years] | 6.2 [0.5 to 34.6] | 6.2 [0.6 to 43.6] | 6.2 [0.5 to 43.6]
Buprenorphine Treatment (years) [Mean (Full Range); unit: years] | 3.5 [0.5 to 10.0] | 3.4 [0.4 to 10.0] | 3.5 [0.4 to 10.0]
Highest Dose of Buprenorphine Treatment Ever Taken (mg/day) [Mean (Inter-Quartile Range); unit: mg/day] | 14 [2.0 to 32.0] | 14 [4.0 to 36.0] | 14 [2.0 to 36.0]
Dose of BPN treatment prior to randomization. [Count of Participants; unit: Participants]
  2 mg/d | 6 | 3 | 9
  4 mg/d | 12 | 15 | 27
  6 mg/d | 8 | 4 | 12
  8 mg/d | 61 | 67 | 128

OUTCOME MEASURES:

1. Primary Outcome: The Primary Efficacy Endpoint is a Responder Rate Analysis, Where a Responder is Defined as a Patient With no More Than 2 of 6 Months With Any Evidence of Illicit Opioid Use.
Description: The primary efficacy endpoint is a responder analysis. A subject will be designated as a responder (meaning they have maintained stability) if they have no more than 2 of 6 months with any evidence of illicit opioid use. Evidence of illicit opioid use is defined as a positive opioid urine toxicology result or self-reported illicit opioid use.
Time Frame: 24 weeks
Population: The analyses included 173 subjects in the ITT population who received treatment and post-baseline evaluations.
Measure: Count of Participants; unit: Participants
Arm/Group | Buprenorphine Implants + Placebo Tablets | Buprenorphine Tablets + Placebo Implants
Number analyzed (Participants) | 84 | 89
Participants
  Responder | 81 | 78
  Non-Responder | 3 | 11
Statistical Analysis 1: Comparison: Buprenorphine Implants + Placebo Tablets vs Buprenorphine Tablets + Placebo Implants; Test type: Non-Inferiority — For the primary efficacy variable, a test of non-inferiority of Probuphine (active) versus SL BPN (control) responders was conducted. A non-inferiority margin of 20% was employed to define noninferiority. A Confidence Interval (CI) for the difference in proportions was calculated, and non-inferiority was established if the lower bound of the 95% CI for the difference of proportions (Probuphine - SL BPN) was greater than -0.20; p < .001, Chi-squared; Difference in Response Rate = 0.088, 95% CI 2-sided [0.009 to 0.167]

2. Secondary Outcome: Percent of Subjects With no Urine Illicit Opioid Use by Month;
Description: The secondary outcome is the percent of subjects with no urine illicit opioid use by month.
Time Frame: 24 weeks
Population: Outcome measures were obtained for all subjects as described in the Analysis Population Description of the primary outcome above.
Measure: Count of Participants; unit: Participants
Arm/Group | Buprenorphine Implants + Placebo Tablets | Buprenorphine Tablets + Placebo Implants
Number analyzed (Participants) | 84 | 89
Participants
  Month 1: Yes | 80 | 84
  Month 1: No | 4 | 5
  Month 2: Yes | 80 | 79
  Month 2: No | 4 | 10
  Month 3: Yes | 83 | 78
  Month 3: No | 1 | 11
  Month 4: Yes | 80 | 80
  Month 4: No | 4 | 9
  Month 5: Yes | 81 | 79
  Month 5: No | 3 | 10
  Month 6: Yes | 76 | 76
  Month 6: No | 8 | 13
Statistical Analysis 1: Comparison: Buprenorphine Implants + Placebo Tablets vs Buprenorphine Tablets + Placebo Implants; Test type: Superiority — At month 6 comparing those subject with no illicit drug use; p = 0.306, Chi-squared

3. Secondary Outcome: Number of Participants With Evidence of Urine Illicit Opioid Use by Month
Description: Secondary efficacy endpoint measures number of participants with evidence of urine illicit opioid use by month.
Time Frame: 24 weeks
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Buprenorphine Implants + Placebo Tablets | Buprenorphine Tablets + Placebo Implants
Number analyzed (Participants) | 84 | 89
Participants
  Month 1: Yes | 4 | 5
  Month 1: No | 80 | 84
  Month 2: Yes | 7 | 12
  Month 2: No | 77 | 77
  Month 3: Yes | 7 | 21
  Month 3: No | 77 | 68
  Month 4: Yes | 8 | 22
  Month 4: No | 76 | 67
  Month 5: Yes | 8 | 22
  Month 5: No | 76 | 67
  Month 6: Yes | 12 | 25
  Month 6: No | 72 | 64
Statistical Analysis 1: Comparison: Buprenorphine Implants + Placebo Tablets vs Buprenorphine Tablets + Placebo Implants; Test type: Superiority; p = .037, Log Rank

4. Secondary Outcome: Percent of Subjects With no Self-reported Illicit Drug Use by Month
Description: Subjects in the ITT population with no self-reported use of any illicit drugs (opioid or non-opioid) by month of evaluation
Time Frame: 24 weeks
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Buprenorphine Implants + Placebo Tablets | Buprenorphine Tablets + Placebo Implants
Number analyzed (Participants) | 84 | 89
Participants
  Week 4: Yes | 72 | 75
  Week 4: No | 12 | 14
  Week 8: number analyzed (Participants) | 83 | 89
  Week 8: Yes | 70 | 75
  Week 8: No | 13 | 14
  Week 12: number analyzed (Participants) | 83 | 88
  Week 12: Yes | 75 | 71
  Week 12: No | 8 | 17
  Weeek 16: number analyzed (Participants) | 81 | 88
  Weeek 16: Yes | 68 | 74
  Weeek 16: No | 13 | 14
  Week 20: number analyzed (Participants) | 81 | 86
  Week 20: Yes | 70 | 70
  Week 20: No | 11 | 16
  Week 24/EOT: number analyzed (Participants) | 81 | 86
  Week 24/EOT: Yes | 68 | 68
  Week 24/EOT: No | 13 | 18

5. Secondary Outcome: Measures of Craving: Desire to Use Visual Analogue Scale (VAS)
Description: The secondary outcome of measures of craving: desire to use is a change from Day 1 (baseline) in the unipolar visual analogue scale (VAS), which is a 0-100 mm scale, where 0 mm is no desire, and 100 mm is strongest possible desire.
Time Frame: 24 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Buprenorphine Implants + Placebo Tablets | Buprenorphine Tablets + Placebo Implants
Number analyzed (Participants) | 84 | 89
units on a scale
  Day 1 (Baseline) | 5.4 (13.98) | 6.8 (16.02)
  Week 4(Change from BL) | 1.1 (17.69) | -1.5 (13.93)
  Week 8(Change from BL) | -1.8 (10.63) | -2.2 (16.38)
  Week 12(Change from BL) | -2.0 (9.37) | -2.2 (16.38)
  Week 16(Change from BL) | -2.2 (11.88) | -2.3 (17.36)
  Week 20(Change from BL) | -2.3 (10.94) | -3.8 (16.17)
  Week 24(Change from BL) | -2.3 (11.15) | -2.8 (19.57)
Statistical Analysis 1: Comparison: Buprenorphine Implants + Placebo Tablets vs Buprenorphine Tablets + Placebo Implants; Comparing change in baseline to week 24 between the two groups; Test type: Superiority; p = 0.832, ANOVA; Mean Difference (Final Values) = -0.4

6. Secondary Outcome: Measures of Withdrawal: Clinical Opiate Withdrawal Scale (COWS)
Description: The secondary outcome measures the change in baseline in the Clinical opiate withdrawal scale (COWS), which is a scale consisting of 11 common opiate withdrawal signs or symptoms, rated on a numeric scale with higher scores associated with greater withdrawal symptoms. A total score was calculated as the sum of the responses to the 11 signs/symptoms for a total range of 0-48. Withdrawal severity was classified, based on the total score, as follows: 0-4=none/normal, 5-12=mild, 13-24=moderate, 25-36=moderately severe, more than 36=severe withdrawal.
Time Frame: 24 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Buprenorphine Implants + Placebo Tablets | Buprenorphine Tablets + Placebo Implants
Number analyzed (Participants) | 84 | 89
units on a scale
  Day 1 (Baseline) | 5.4 (15.18) | 6.0 (13.02)
  Week 4(Change from BL) | -0.8 (12.70) | -1.2 (16.91)
  Week 8(Change from BL) | -2.0 (11.45) | -1.9 (16.38)
  Week 12(Change from BL) | -2.3 (11.12) | -2.4 (14.72)
  Week 16(Change from BL) | -2.4 (15.36) | -2.3 (15.39)
  Week 20(Change from BL) | -2.8 (12.03) | -3.4 (13.79)
  Week 24(Change from BL) | -2.7 (12.58) | -1.9 (18.97)
Statistical Analysis 1: Comparison: Buprenorphine Implants + Placebo Tablets vs Buprenorphine Tablets + Placebo Implants; Test type: Superiority; p = 0.922, ANOVA; Mean Difference (Final Values) = -0.0

7. Secondary Outcome: Measures of Withdrawal: Subjective Opioid Withdrawal Scale (SOWS) (ITT Population)
Description: The secondary outcome measures the change in baseline in the subjective opioid withdrawal scale (SOWS), which is a scale which is a subject self-assessment of withdrawal symptoms. The scale consists of 16 questions that rate the intensity of withdrawal from 0 (not at all) to 4 (extremely) with a cumulative score ranging from 0-64 (0 =not at all, 64=extremely)
Time Frame: 24 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Buprenorphine Implants + Placebo Tablets | Buprenorphine Tablets + Placebo Implants
Number analyzed (Participants) | 84 | 89
units on a scale
  Day 1 (Baseline) | 2.7 (3.85) | 2.2 (3.15)
  Week 4 (Change from BL) | 0.3 (55.56) | 0.3 (5.51)
  Week 8(Change from BL) | -1.1 (3.39) | 0.4 (5.63)
  Week 12(Change from BL) | -0.4 (5.53) | -0.1 (4.15)
  Week 16(Change from BL) | -0.2 (5.23) | -0.4 (4.25)
  Week 20(Change from BL) | -0.9 (4.47) | -0.1 (4.47)
  Week 24(Change from BL) | 0.1 (5.26) | 0.1 (5.26)
Statistical Analysis 1: Comparison: Buprenorphine Implants + Placebo Tablets vs Buprenorphine Tablets + Placebo Implants; Test type: Superiority; p = 0.425, ANOVA; Mean Difference (Final Values) = -0.6

8. Secondary Outcome: Measures of Craving: Need to Use Visual Analogue Scale (VAS)
Description: The secondary outcome of measures of craving: Need to use is a change from Day 1 (baseline) in the unipolar visual analogue scale (VAS), which is a 0-100 mm scale, where 0 mm is no need, and 100 mm is strongest possible need.
Time Frame: 24 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Buprenorphine Implants + Placebo Tablets | Buprenorphine Tablets + Placebo Implants
Number analyzed (Participants) | 84 | 89
units on a scale
  Day 1 (Baseline): number analyzed (Participants) | 83 | 89
  Day 1 (Baseline) | 5.4 (15.18) | 6.0 (13.02)
  Week 4(Change from BL): number analyzed (Participants) | 83 | 89
  Week 4(Change from BL) | -0.8 (12.70) | -1.2 (16.91)
  Week 8(Change from BL): number analyzed (Participants) | 83 | 89
  Week 8(Change from BL) | -2.0 (11.45) | -1.9 (16.93)
  Week 12(Change from BL): number analyzed (Participants) | 83 | 89
  Week 12(Change from BL) | -2.3 (11.12) | -2.4 (14.72)
  Week 16(Change from BL): number analyzed (Participants) | 83 | 89
  Week 16(Change from BL) | -2.4 (15.36) | -2.3 (15.39)
  Week 20(Change from BL): number analyzed (Participants) | 83 | 89
  Week 20(Change from BL) | -2.8 (12.03) | -3.4 (13.79)
  Week 24(Change from BL): number analyzed (Participants) | 83 | 89
  Week 24(Change from BL) | -2.7 (12.58) | -1.9 (18.97)
Statistical Analysis 1: Comparison: Buprenorphine Implants + Placebo Tablets vs Buprenorphine Tablets + Placebo Implants; Comparing change in baseline to week 24 between the two groups; Test type: Superiority; p = 0.505, ANOVA; Median Difference (Final Values) = -1.3

ADVERSE EVENTS:
Time Frame: All AEs were documented and followed from the time the subject signed the ICF until 14 days after the EOT Visit (i.e., implant removal and discontinuation of SL BPN/placebo treatment) which was approximately 28 weeks. Serious adverse events and AEs designated as possibly related to study drug were followed until resolution or stabilization.
Description: For the purpose of this report, AEs considered by the investigator to be possibly, probably, or definitely related to study drug are classified as study drug-related events.
Arm/Group | Buprenorphine Implants + Placebo Tablets | Buprenorphine Tablets + Placebo Implants
Serious Adverse Events (participants affected / at risk) | 2/87 | 3/89
Other Adverse Events (participants affected / at risk) | 1/87 | 4/89
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Buprenorphine Implants + Placebo Tablets (N=87) | Buprenorphine Tablets + Placebo Implants (N=89)
Biliary Colic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 1 (1) | 0 (0)
Bipolar I Disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Cholecystitis Chronic (Hepatobiliary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1.15% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Buprenorphine Implants + Placebo Tablets (N=87) | Buprenorphine Tablets + Placebo Implants (N=89)
Muscle spasm (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Abortion - Spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Pediatric exposure to treatment (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Cellulitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No